CLINICAL TRIAL: NCT01994109
Title: A Phase 3, Multicenter, Double-Blind, Placebo-Controlled, Single-Treatment Efficacy and Safety Study of MYOBLOC® (Part A) Followed by Open-Label, Multiple-Treatment With MYOBLOC® (Part B) in the Treatment of Troublesome Sialorrhea in Adult Subjects
Brief Title: Efficacy and Safety Study of MYOBLOC® Followed by Open-Label Multiple-Treatment With MYOBLOC® in the Treatment of Troublesome Sialorrhea in Adult Subjects
Acronym: MYSTICOL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Supernus Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SN-SIAL-301
Record Dates: First submitted 2013-11-14; First posted 2013-11-25 (Estimated); Results first posted 2019-08-15 (Actual); Last update posted 2021-07-13 (Actual); Status verified 2019-08

CONDITIONS: Sialorrhea
Keywords: Sialorrhea; Parkinson's disease; Amyotrophic lateral sclerosis (ALS); stroke; neuroleptics
MeSH Terms: conditions — Sialorrhea; Parkinson Disease; Amyotrophic Lateral Sclerosis; Stroke | interventions — rimabotulinumtoxinB

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- MYOBLOC 2500 U (Active Comparator): Subjects will receive specified dose of MYOBLOC
  Interventions: Drug: MYOBLOC
- MYOBLOC 3500 U (Active Comparator): Subjects will receive specified dose of MYOBLOC
  Interventions: Drug: MYOBLOC
- Placebo (Placebo Comparator): Subjects will receive volume matched Placebo
  Interventions: Other: PLACEBO

INTERVENTIONS:
Drug: MYOBLOC — MYOBLOC (rimabotulinumtoxinB) Injection, or botulinum toxin type B, is the "B" serotype of botulinum toxin. It is the only commercially available "B" serotype, and also the only available botulinum toxin that does not require reconstitution for use.
  Other Names: rimabotulinumtoxinB, botulinum toxin type B
  Arms: MYOBLOC 2500 U; MYOBLOC 3500 U
Other: PLACEBO
  Other Names: volume-matched placebo
  Arms: Placebo

SUMMARY:
This study will evaluate the efficacy and safety of MYOBLOC in the treatment of Sialorrhea (drooling), which can be a symptom of many disease conditions. MYOBLOC will be injected directly into the salivary glands. MYOBLOC has been shown in previous trials to safely decrease saliva production, thereby demonstrating its potential as a safe and effective treatment for troublesome sialorrhea.

ELIGIBILITY:
Inclusion Criteria:

* Seeking treatment for troublesome sialorrhea for at least 3 months that is occurring secondary to any disorder or related to any cause
* Investigator sites will review entire list of inclusion criteria with potential subjects

Exclusion Criteria:

* Any known prior exposure to botulinum toxin type B, or known adverse reaction or sensitivity to botulinum toxin type A, or known sensitivity to any of the MYOBLOC solution components.
* Prior botulinum toxin treatment to the salivary glands at any time
* Investigator sites will review entire list of exclusion criteria with potential subjects

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 187 (Actual)
Dates: Start 2013-11; Primary Completion 2016-01 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Najeebah Abdul-Musawir, MD,MBA, Study Director — Supernus Pharmaceuticals, Inc.
Locations (34):
- United States (24):
  - Loma Linda, California
  - Los Angeles, California
  - National City, California
  - Aurora, Colorado
  - Washington D.C., District of Columbia
  - Boca Raton, Florida
  - Port Charlotte, Florida
  - Carmel, Indiana
  - Baltimore, Maryland
  - Elkridge, Maryland
  - Detroit, Michigan
  - St Louis, Missouri
  - Edison, New Jersey
  - Albany, New York
  - New York, New York
  - Cincinnati, Ohio
  - Tulsa, Oklahoma
  - Port Royal, South Carolina
  - Cordova, Tennessee
  - Houston, Texas
  - San Antonio, Texas
  - Salt Lake City, Utah
  - Kirkland, Washington
  - Tacoma, Washington
- Russia (4):
  - Irkutsk, Irkutsk Oblast
  - Vsevolozhsk, Leningradskaya Oblast'
  - Saint Petersburg, Petrodvorets
  - Krasnoyarsk
- Ukraine (6):
  - Dnipropetrovsk
  - Ivano-Frankivsk
  - Kharkiv
  - Lviv
  - Rivne
  - Uzhhorod

REFERENCES:
- [Result] Chinnapongse R, Gullo K, Nemeth P, Zhang Y, Griggs L. Safety and efficacy of botulinum toxin type B for treatment of sialorrhea in Parkinson's disease: a prospective double-blind trial. Mov Disord. 2012 Feb;27(2):219-26. doi: 10.1002/mds.23929. Epub 2011 Sep 1. PMID 21887710
- [Result] Ondo WG, Hunter C, Moore W. A double-blind placebo-controlled trial of botulinum toxin B for sialorrhea in Parkinson's disease. Neurology. 2004 Jan 13;62(1):37-40. doi: 10.1212/01.wnl.0000101713.81253.4c. PMID 14718694
- [Derived] Isaacson SH, Ondo W, Jackson CE, Trosch RM, Molho E, Pagan F, Lew M, Dashtipour K, Clinch T, Espay AJ; MYSTICOL Study Group. Safety and Efficacy of RimabotulinumtoxinB for Treatment of Sialorrhea in Adults: A Randomized Clinical Trial. JAMA Neurol. 2020 Apr 1;77(4):461-469. doi: 10.1001/jamaneurol.2019.4565. PMID 31930364

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 33 sites including United States, Russia and Ukraine.
Pre-assignment Details: DB: Double Blind (Part A) OL: Open Label (Part B)
Groups:
- DB: MYOBLOC 2500 U; DB: MYOBLOC 3500 U: Participants will receive specified dose of MYOBLOC
- DB: Placebo: Participants will receive volume matched Placebo
- OL: ALL MYOBLOC: All Participants were to receive 3500 U MYOBLOC but could receive lower doses at investigator discretion.
Period: Double-blind Phase (Part A)
Arm/Group | DB: MYOBLOC 2500 U | DB: MYOBLOC 3500 U | DB: Placebo | OL: ALL MYOBLOC
Started | 63 | 64 | 60 | 0
Completed | 62 | 61 | 53 | 0
Not Completed | 1 | 3 | 7 | 0
Period: Open-label Phase (Part B)
Arm/Group | DB: MYOBLOC 2500 U | DB: MYOBLOC 3500 U | DB: Placebo | OL: ALL MYOBLOC
Started | 0 | 0 | 0 (No placebo group in Part B.) | 170 (61 from 2500 U group, 57 from 3500 U group, 52 from Placebo group continued to Part B)
Completed | 0 | 0 | 0 (No placebo group in Part B.) | 128
Not Completed | 0 | 0 | 0 | 42

BASELINE CHARACTERISTICS:
Population: Demographic Characteristics of intent-to-treat (ITT) Population.
Groups:
- MYOBLOC 2500 U: Subjects were dosed per treatment assignment of 2500 U MYOBLOC.
- MYOBLOC 3500 U: Subjects were dosed per treatment assignment of 3500 U MYOBLOC.
- PLACEBO: Placebo was dosed as an exact match of MYOBLOC.
- Total: Total of all reporting groups
Arm/Group | MYOBLOC 2500 U | MYOBLOC 3500 U | PLACEBO | Total
Number analyzed (Participants) | 63 | 64 | 57 | 184
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 29 | 25 | 24 | 78
  >=65 years | 34 | 39 | 33 | 106
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.6 (13.0) | 64.6 (14.0) | 64.1 (13.1) | 63.8 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 9 | 16 | 40
  Male | 48 | 55 | 41 | 144
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 2 | 1 | 8
  Not Hispanic or Latino | 58 | 62 | 56 | 176
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 1 | 0 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 1 | 1 | 4
  White | 60 | 60 | 55 | 175
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Unstimulated Salivary Flow Rate (USFR) at Week 4 Post-injection Visit (Part A)
Description: Change weight of expectorated saliva at a Week 4 post-injection visit.
Time Frame: 4 Weeks
Population: The per protocol included subjects with a minimum USFR of 0.2 g/min.
Measure: Least Squares Mean (Standard Error); unit: g/minute
Arm/Group | MYOBLOC 2500 U | MYOBLOC 3500 U | Placebo
Number analyzed (Participants) | 63 | 64 | 57
g/minute | -0.37 (0.03) | -0.36 (0.03) | -0.07 (0.03)
Statistical Analysis 1: Comparison: MYOBLOC 3500 U vs Placebo; Test type: Superiority; p < 0.0001, ANCOVA
Statistical Analysis 2: Comparison: MYOBLOC 2500 U vs Placebo; Test type: Superiority; p < 0.0001, ANCOVA

2. Primary Outcome: Clinical Global Impression Change (CGI-C) at Week 4 Post-injection (Part A)
Description: CGI-C was assessed on a 7-point scale ranging from "very much improved" to "very much worse" with 1 assigned to "very much improved" and 7 assigned to "very much worse"; ranging from a minimum score of 1 and a maximum score of 7.
Time Frame: 4 weeks
Population: Per protocol the intent-to-treat population who were injected with study medication and had at least 1 post injection CGI-C measurement up to week 4 (inclusive).
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | MYOBLOC 2500 U | MYOBLOC 3500 U | Placebo
Number analyzed (Participants) | 63 | 64 | 60
score on a scale | 2.38 (0.12) | 2.45 (0.12) | 3.59 (0.13)
Statistical Analysis 1: Comparison: MYOBLOC 3500 U vs Placebo; Test type: Superiority; p < 0.0001, ANCOVA
Statistical Analysis 2: Comparison: MYOBLOC 2500 U vs Placebo; Test type: Superiority; p < 0.0001, ANCOVA

ADVERSE EVENTS:
Time Frame: Part A: 13-Week Post-Injection Period; Part B: 4 Sessions of 13-Week (+/- 2 Weeks) Post-Injection Periods
Description: Part A (Session 1): Serious TEAEs Reported During Double-Blind Phase (Safety Population) Part B (Sessions 2-5): Serious TEAEs Reported During Open-Label Phase (OL Population)
Groups:
- MYOBLOC 2500 U (Part A); MYOBLOC 3500 U (Part A): Participants received specified dose of MYOBLOC. Participants were evaluated for 13 weeks following the injection.
- Placebo (Part A): Participants received volume matched Placebo. Participants were evaluated for 13 weeks following the injection.
- OL: ALL MYOBLOC (Part B): Participants received Open Label treatment with 3500 U (decreased dose at investigator discretion) every 13 weeks for a maximum of 4 treatment sessions.
Arm/Group | MYOBLOC 2500 U (Part A) | MYOBLOC 3500 U (Part A) | Placebo (Part A) | OL: ALL MYOBLOC (Part B)
All-Cause Mortality (participants affected / at risk) | 0/63 | 2/64 | 1/60 | 9/170
Serious Adverse Events (participants affected / at risk) | 1/63 | 4/64 | 4/60 | 32/170
Other Adverse Events (participants affected / at risk) | 44/63 | 38/64 | 16/60 | 143/170
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MYOBLOC 2500 U (Part A) (N=63) | MYOBLOC 3500 U (Part A) (N=64) | Placebo (Part A) (N=60) | OL: ALL MYOBLOC (Part B) (N=170)
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1 | 0 | 2
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Malaise (General disorders) | 0 | 1 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 5
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 3
Urosepsis (Infections and infestations) | 0 | 0 | 1 | 0
Brain cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Nodular melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 2
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Circulatory collapse (Vascular disorders) | 0 | 0 | 1 | 0
Atrial fibrillaiton (Cardiac disorders) | 0 | 0 | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 1
Visual acuity reduced (Eye disorders) | 0 | 0 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Asthenia (General disorders) | 0 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 0 | 1
Hypothermia (General disorders) | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1
Fungal skin infection (Infections and infestations) | 0 | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1
Staphylococcal infection (Infections and infestations) | 0 | 0 | 0 | 1
Burns first degree (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Burns second degree (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Pharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Amyotrophic lateral sclerosis (Nervous system disorders) | 0 | 0 | 0 | 1
Dementia with Lewy bodies (Nervous system disorders) | 0 | 0 | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 2
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 0 | 1
Parkinson's disease (Nervous system disorders) | 0 | 0 | 0 | 1
Parkinsonism (Nervous system disorders) | 0 | 0 | 0 | 1
Radiculopathy (Nervous system disorders) | 0 | 0 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 1
Vocal cord paralysis (Nervous system disorders) | 0 | 0 | 0 | 1
Aggression (Psychiatric disorders) | 0 | 0 | 0 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 3
Arteriosclerosis (Vascular disorders) | 0 | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MYOBLOC 2500 U (Part A) (N=63) | MYOBLOC 3500 U (Part A) (N=64) | Placebo (Part A) (N=60) | OL: ALL MYOBLOC (Part B) (N=170)
Dental caries (Gastrointestinal disorders) | 5 | 3 | 2 | 50
Dry mouth (Gastrointestinal disorders) | 24 | 29 | 5 | 73
Dysphagia (Gastrointestinal disorders) | 7 | 3 | 1 | 21
Fall (Injury, poisoning and procedural complications) | 4 | 3 | 4 | 28
Dizziness (Nervous system disorders) | 4 | 0 | 0 | 10
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 4 | 8
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 12
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 11
Weight decreased (Investigations) | 0 | 0 | 0 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the first right, within 9 months following the later to occur 1) close out meeting or 2) Sponsor possessing all data, to publish the lead paper. Following the foregoing, Institution has the right to publish the results provided the Institution provides a Publications Committee, which includes the Sponsor, with a draft at least 30 days before submission. At Sponsor's request, Institution shall withhold publication for 45 days to allow filing of a patent application.